CLINICAL TRIAL: NCT01929473
Title: Seroepidemiological Study of Pertussis and Other Infectious Diseases
Status: Completed | Type: Observational
Sponsor: Gifu Prefecture Medical Association (Other)
Collaborators: Sanofi Pasteur S.A. (Unknown)
Responsible Party: Sponsor
Other Study IDs: G-P001
Record Dates: First submitted 2013-08-15; First posted 2013-08-28 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Pertussis Infection
Keywords: Pertussis infection; Risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Serum samples will be corrected twice from the same youth subjects with one year interval.

Seroincidence of pertussis will be estimated by the elevation of Ig-G-PT in paired sera from an identical individual.

The relationship between the incidence and the demographic data or medical history of the subjects will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Students of junior high school, high schools or college in Gifu prefecture
* Students who can have the second blood drawing one year later
* Students (and their parent when students are underage) whose written consent is obtainable.

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students of junior high school, high school or college
Sampling Method: Probability Sample
Enrollment: 3830 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Kawai, Study Chair — Gifu Prefecture Medial Association
Locations (1):
- Gifu, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood Drawings (0 Day, 365 Day) and Questionnaires
Started | 3830 (0 day)
365 Day | 3589
Completed | 3243
Not Completed | 587

BASELINE CHARACTERISTICS:
Arm/Group | Blood Drawings (0 Day, 365 Day) and Questionnaires
Number analyzed (Participants) | 3243
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1605
  Male | 1638
Region of Enrollment [Number; unit: participants]
  Japan | 3243

OUTCOME MEASURES:

1. Primary Outcome: IgG
Description: Seroincidence of pertussis estimated by the elevation of Ig-G-PT in paired sera(0day, 365day).
Time Frame: 0 day, 365 day (2 points)
Measure: Mean (Standard Deviation); unit: EU/mL(log transformed)
Arm/Group | Blood Drawings (0 Day, 365 Day) and Questionnaires
Number analyzed (Participants) | 3243
EU/mL(log transformed)
  0 day | 1.254 (0.008)
  365 day | 1.258 (0.007)

2. Secondary Outcome: Incidence of Pertussis
Description: Questionnaire
Time Frame: 0 day
Reporting Status: Not Posted

3. Secondary Outcome: Antibodies of Varicella, Mumps and Rubella
Description: Questionnaire
Time Frame: 0 day
Reporting Status: Not Posted

4. Secondary Outcome: Infection Risk Factors Including Family Numbers, Living Space, With or Without a Cough Patient in the Surroundings, Medical History and Hospitalization
Description: Questionnaire
Time Frame: 365 day
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Blood Drawings (0 Day, 365 Day) and Questionnaires
Serious Adverse Events (participants affected / at risk) | 0/3243
Other Adverse Events (participants affected / at risk) | 0/3243

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other